CLINICAL TRIAL: NCT02128503
Title: Prevalence and Clinical Course of Chronic Hepatitis B Infection in Patients With Inflammatory Bowel Disease and Rheumatologic Disease on Immunosuppressive Therapy
Brief Title: Prevalence and Clinical Course of Chronic Hep B Infection in IBD and Rheumatologic Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sample size recruited is not enough
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IBD-RA HBV
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Inflammatory Bowel Disease; Crohn Disease; Ulcerative Colitis; Rheumatic Diseases; Hepatitis B, Chronic
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Rheumatic Diseases; Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HBV DNA level monitoring (Other): Group with HBV DNV level being monitored regularly
  Interventions: Other: HBV DNA level monitoring

INTERVENTIONS:
Other: HBV DNA level monitoring — HBV DNV level being monitoring regularly

SUMMARY:
This study aims to determine the prevalence of HBV infection in patients with IBD and rheumatologic disease, and to assess the impact of immunosuppressive therapy on viral load and clinical course of IBD patients.

DETAILED DESCRIPTION:
The incidence of inflammatory bowel disease (IBD) has been increasing in Hong Kong. The management of inflammatory bowel disease involved the use of immunosuppressant, however, the use of immunosuppressant in patients with hepatitis B infection has been associated with hepatitis B reactivation. It is estimated that around 7% of the Hong Kong population is infected with HBV. The information on the prevalence of hepatitis B in IBD patients in Hong Kong is lacking. Moreover, limited information is available on the effect of different immunosuppressive regimens given for longer periods of time in lower doses in patients with chronic HBV infection and IBD. There is therefore a need to determine the incidence and predictive factors for HBV reactivation in these patients.

Rheumatologic diseases, including systemic lupus erythematous, rheumatoid arthritis, psoriasis and anklyosing spondylitis are inflammatory conditions which commonly affect the locomotors system as well as other organs. Epidemiological data from China have suggested that patients with ankylosing spondylitis have a higher risk of hepatitis B infection; while the rates of hepatitis B for those with rheumatoid arthritis, and other spondyloathropathies are similar to that of the general population. However, there are no such local data in Hong Kong aspect.

This study aims to determine the prevalence of HBV infection in patients with IBD and rheumatologic disease, and to assess the impact of immunosuppressive therapy on viral load and clinical course of IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* All IBD and rheumatologic patients aged 18 years or older

Exclusion Criteria:

* Lack of consent
* Patients with evidence of other chronic liver disease,metabolic syndrome, men consuming more than 30 g of alcohol per day and women consuming more than 20 g of alcohol per day, patients with liver decompensation, HCC, previous liver surgery or liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-10-16 (Actual); Study Completion 2015-10-16 (Actual)

PRIMARY OUTCOMES:
Changes in HBV DNA levels | 2 Years
  Changes in HBV DNA levels in patients with chronic hepatitis B and IBD treated with immunosuppressants

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No